CLINICAL TRIAL: NCT05518214
Title: 'Oral Microbiome -Dietary Nitrate' Interactions and Cognitive Health in Older Age
Acronym: COGNIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COGNIT
Record Dates: First submitted 2022-07-25; First posted 2022-08-26 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Dietary Supplementations

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind study where both the Participant and Investigator are blind to the supplement given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beetroot (Experimental): Participants will receive nitrate-rich (70 ml, containing 6.4 mmol of nitrate) beetroot juice, by Beet It, James White. Participants will take 1 beetroot juice drink everyday for 12 weeks.
  Interventions: Dietary Supplement: Beetroot
- Placebo (Placebo Comparator): Participants will receive a placebo beetroot juice with the nitrate removed, by Beet It, James White. Participants will take 1 placebo juice drink everyday for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot — Participants receive a 12-week supply of beetroot juice.
  Arms: Beetroot
Dietary Supplement: Placebo — Participants receive a 12-week supply of placebo beetroot juice.
  Arms: Placebo

SUMMARY:
Vegetable rich diets contain natural inorganic nitrate. These diets are linked to good heart and brain health. Human cells cannot 'activate' nitrate. Humans must rely on specific bacteria living in the mouth to digest nitrate to an active form called 'nitric oxide' that we can use in the body. We have found that nitrate makes the oral microbiome healthier and improves nitric oxide production. This study will investigate whether changes in oral bacteria caused by dietary nitrate are linked to any changes in brain performance.We will ask 60 healthy men and women of over 50 years of age to take part. We will ask them to drink either nitrate-rich beetroot juice or placebo juice daily for 12 weeks. We will do this investigation entirely remotely by using online tools and by posting of supplements and samples. We will sample the volunteers' oral microbiome and assess their cognitive performance before and after dietary supplementation. We will analyse the nitric oxide content in the samples that the volunteers post us. We will try to findgroups of bacteria linked with goodbrainfunction.The results will help us better understand how oral bacteria may influence cognitive function in older age.

DETAILED DESCRIPTION:
Oral dysbiosis and poor dental health have been associated with impaired cardiovascular and cognitive health, but it is not known which characteristics of bacterial communities specifically might mediate such relationships. One mechanism by which the oral microbiota may influence health is its contribution to production of the signalling molecule, nitric oxide (NO), which, among many other functions, regulates vascular tone and neurotransmission . The capacity for endogenous NO production via the enzymatic NOS synthase pathway declines in older age, contributing to development of arterial hypertension, reduced physical and cognitive functional capacity, and increased morbidity. Therefore, the composition of the oral microbiota may be particularly important to enable older people to benefit from a nitrate-rich diets, such as the Mediterranean diet, which has been associated with reduced risk of developing dementia in older age. A key genetic risk factor for dementia is a form of apolipoprotein E gene called APOE4, which may also modulate responsiveness to dietary interventions.The purpose of this research is to investigate whether specific groups of oral bacteria, that are sensitive to change with dietary nitrate supplementation, are correlated with indices of cognitive function (primary objective) as well as APOE genotype, diet, physical activity, and markers of vascular health (secondary objectives), in people over 50 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent.
* Male or Female.
* Over 50 years of age.
* Access to a postal service (Royal Mail)
* Access to the Internet.
* Mainland UK resident.
* APOE genotype available in PROTECT database.

Exclusion Criteria:

* Diagnosis of dementia, because the participant may be unable to provide informed consent.
* Current or previous smoker (within the last year).
* Regular drinkers of alcoholic beverages which are over 14% ABV undiluted.
* Current or recent use of antibiotics (within the past 3 months).
* Self-reported substantial use of mouthwash or tongue scrapers within the past month.
* Self-reported periodontitis, gingivitis or other oral disease.
* No available APOE genotyping in PROTECT database.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline oral bacteria co-occurrence at 12 weeks using oral microbiome abundance data and WGCNA analysis. | Change measured between baseline and 12-weeks post-intervention.
  Identify co-occurring clusters of oral bacteria which are consistently related to indices of cognitive status across dietary interventions with nitrate and placebo. Using oral microbiome abundance data from sequenced oral microbiome DNA in the mouth rinse samples, the change from baseline to post-12 week intervention is measured. WGCNA analysis is used to cluster co-occurring bacteria and detect patterns of grouping.

SECONDARY OUTCOMES:
Change from baseline oral nitric oxide bioavailability at 12 weeks using ozone-based chemiluminescence. | Change measured between baseline and 12-weeks post-intervention.
  The change from baseline to post-12 week intervention nitrate and nitrite concentrations in mouth rinse samples is measured using ozone-based chemiluminescence.
Change from baseline composition of the oral microbiome at 12 weeks using oral microbiome abundance data from sequencing oral microbiome DNA in mouth rinse samples. | Change measured between baseline and 12-weeks post-intervention.
  Oral microbiome sequencing of bacterial DNA isolated from mouth rinse samples. The change in the composition of the oral microbiome is measured from baseline to post-12 week intervention using oral microbiome abundance data.
Change from baseline cognitive status at 12 weeks. | Change measured between baseline and 12-weeks post-intervention.
  'Factors of Longitudinal Attention, Memory and Executive Function' (FLAME) composite score. Online FLAME cognitive assessment battery completed at home by the participants via the online PROTECT study. The FLAME cognitive assessment is a validated battery of online cognitive tests where correct/incorrect responses and response time are measured.
Correlation between oral microbiome and existing descriptive data. | Correlation measured after 12-weeks post-intervention.
  Correlation of oral microbiome with existing PROTECT cohort variables (APOE genotype, diet, physical activity). The oral microbiome abundance data is correlated with APOE genotype and dietary and physical questionnaire data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter Sport and Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briskey D, Tucker PS, Johnson DW, Coombes JS. Microbiota and the nitrogen cycle: Implications in the development and progression of CVD and CKD. Nitric Oxide. 2016 Jul 1;57:64-70. doi: 10.1016/j.niox.2016.05.002. Epub 2016 May 7. PMID 27164294
- [Background] Stamler JS, Meissner G. Physiology of nitric oxide in skeletal muscle. Physiol Rev. 2001 Jan;81(1):209-237. doi: 10.1152/physrev.2001.81.1.209. PMID 11152758
- [Background] Bryan NS, Tribble G, Angelov N. Oral Microbiome and Nitric Oxide: the Missing Link in the Management of Blood Pressure. Curr Hypertens Rep. 2017 Apr;19(4):33. doi: 10.1007/s11906-017-0725-2. PMID 28353075
- [Background] Vanhatalo A, L'Heureux JE, Kelly J, Blackwell JR, Wylie LJ, Fulford J, Winyard PG, Williams DW, van der Giezen M, Jones AM. Network analysis of nitrate-sensitive oral microbiome reveals interactions with cognitive function and cardiovascular health across dietary interventions. Redox Biol. 2021 May;41:101933. doi: 10.1016/j.redox.2021.101933. Epub 2021 Mar 5. PMID 33721836
- [Background] Brooker H, Williams G, Hampshire A, Corbett A, Aarsland D, Cummings J, Molinuevo JL, Atri A, Ismail Z, Creese B, Fladby T, Thim-Hansen C, Wesnes K, Ballard C. FLAME: A computerized neuropsychological composite for trials in early dementia. Alzheimers Dement (Amst). 2020 Oct 14;12(1):e12098. doi: 10.1002/dad2.12098. eCollection 2020. PMID 33088895